CLINICAL TRIAL: NCT06650800
Title: Effect of Psilocybin on the Positive Valence System in Treatment-resistant Depression: a Pilot Clinical Neuroimaging Study
Brief Title: Effect of Psilocybin on the Positive Valence System in Treatment-resistant Depression
Acronym: PSILODAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NIMAO/2021-2/JLC-01
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Depressive Disorder; Depressive Disorder, Treatment-Resistant; Hallucinogens; Reinforcement, Psychology
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Treatment-Resistant | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient with major depressive episode (Experimental)
  Interventions: Drug: Psilocybin; Other: MRI

INTERVENTIONS:
Drug: Psilocybin — Single-dose psilocybin administration: oral ingestion of one 25 mg capsule
Other: MRI — 1.5 hour brain MRI before and after psilocybin administration

SUMMARY:
The study hypothesis is that the antidepressant effect of psilocybin is mediated by a normalization of the functioning of the positive valence system. Depressive states, especially moderate to severe depressions that associate a certain level of anhedonia, produce an overvaluation of the cost of efforts and an infra-evaluation of the possible rewards derived from an action. Psilocybin would reduce anhedonia and the cost of efforts, facilitating the anticipation of reward. Thus, the antidepressant effect of psilocybin would be mediated by a greater anticipation of rewards (reduction of anhedonia) and a more optimistic estimation of the results of efforts (increase in motivation). Psilocybin-induced changes in the positive valence system will be observable on brain MRI images, particularly in the effort evaluation circuits: basolateral amygdala, dorsal anterior cingulate cortex, ventral pallidum, ventral striatum (VS), ventral tegmental area (VTA). The mesolimbic circuit (VS, VTA) is the anatomical substrate of anticipation of rewarding stimuli (food, sex, drugs). The amygdala also fulfills an associative function between environmental cues and rewarding stimuli. Structural and functional alterations in this circuit are associated with depressive symptoms such as anhedonia or distortions in the perception and memories of rewards. This hypothesis will be tested on a population of patients with moderate or severe depressive symptoms who meet the criteria for TRD.

DETAILED DESCRIPTION:
Depressive disorders are strongly associated with suicide risk and are the leading cause of disability in the world. Psilocybin is a natural alkaloid with psychedelic and hallucinogenic effects, produced by its active metabolite: psilocin. In recent years, there has been a resurgence of research aimed at using psilocybin in the treatment of psychiatric disorders, and in particular depression, combined or not with various psychotherapeutic programs. Psilocybin-assisted therapy is effective in treating cancer-associated depression and resistant depression. The Federal Drug Administration (FDA) has designated it as a "Breakthrough Therapy" in the treatment of treatment-resistant depression (TRD). Most researchers consider that the antidepressant effects of psilocybin are associated with the activation of the serotonin 5-HT2a receptor, with acute neuromodulation effects that modify the connectivity of cortico-striatal loops, but the mechanisms supporting this effect are unknown. The purpose of this study is to verify whether the antidepressant action of psilocybin is associated with an activation of the brain areas involved in the positive valence system, by comparing the activity of the neural circuits responsible for the evaluation of effort before and after taking psilocybin. The correlations between the activation of brain areas and the depression severity, behavioral activation and anhedonia scores will help establish a link with the response to treatment. Finally, the study authors wish to test the feasibility of a study with psilocybin in a French clinical population.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* Patient with a current DSM-IV diagnosis of moderate or severe major depressive episode (MDE) without psychotic features (based on clinical assessment and confirmed by the MINI interview and the QIDS).
* Patient who has not responded to at least two antidepressant treatments of different classes, administered appropriately in terms of dose and duration, for a moderate to severe major depressive episode.
* Patients receiving antidepressant treatment of the SSRI (Selective Serotonin Reuptake Inhibitors) or SNRI (Serotonin Norepinephrine Reuptake Inhibitors) classes may maintain this treatment for the duration of the trial, without modification • Patient with a score > 10 on the QIDS scale.
* Patient available for a 4-month follow-up.
* Patient able to speak and understand French easily.

Exclusion Criteria:

* The patient is participating in a medical product-based interventional study, or is in a period of exclusion determined by a previous study
* Patient unable to express consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient with allergy, hypersensitivity or other adverse reaction to previous use of psilocybin or other hallucinogens.
* Patient who has used hallucinogenic substances (excluding cannabis) more than 5 times in his/her lifetime or at any time in the last twelve months.
* Patient on medication or illicit substances likely to interfere with the effects of psychedelics (urine analysis and breathalyzer on D0).
* Patient with regular consumption of alcoholic beverages (>20 drinks/week)
* Any other major clinically significant concomitant disease that, in the opinion of the investigator, may interfere with the interpretation of the study results or constitute a risk to the health of the participant, if he or she participates in the study
* Patient with a prolonged QTc interval (interval corrected by the Fridericia formula >450 ms for men and >470 ms for women
* Participant planning to donate sperm within three months of psilocybin administration
* Female participant having sexual intercourse that could result in pregnancy and not agreeing to use a highly effective contraceptive method (combined hormonal contraception (containing estrogen and progestin), contraception associated with inhibition of ovulation, hormonal progestin-only contraception associated with inhibition of ovulation, intrauterine device intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner, and sexual abstinence) throughout their participation in the study and for at least three months after psilocybin administration.
* Positive serum pregnancy test at inclusion for participants of childbearing potential. NB: a urine pregnancy test will also be performed on the day of psilocybin administration.
* Pregnant patient (confirmed by pregnancy test), parturient or breastfeeding, or wishing to become pregnant during their participation in the study
* Active substance dependence according to the MINI questionnaire (excluding tobacco).
* Patient whose psychotropic treatment (anxiolytics, antipsychotics, hypnotics, mood stabilizers) has been modified in the last month.
* Patient on antidepressant treatment other than SSRIs or SNRIs. (Antidepressant treatments other than SSRIs or SNRIs are prohibited in the trial. Patients receiving antidepressant treatment of a different class (MAOIs, tricyclics, tetracyclics), alone or in combination, will not be included in the study).
* Patient suffering from intellectual disability (IQ less than or equal to 75).
* Patient with a history of bipolar disorder, schizophrenia, schizoaffective disorder or psychosis not otherwise specified during life.
* Patient with a family history of schizophrenia, schizoaffective disorder or bipolar disorder type 1 in first or second degree relatives.
* Patient who has started psychotherapy in the 30 days preceding the screening visit, or whose psychotherapy is likely to undergo changes during the clinical trial.
* Patient who has received in the last 6 months treatments such as: ECT, vagus nerve stimulation, deep brain stimulation, transcranial magnetic stimulation.
* Patient with any disease or unstable physical condition determined by clinical examination, history or laboratory tests (ECG, blood test at inclusion) These pathologies include cardiovascular comorbidities: history of stroke, myocardial infarction, heart failure, intracranial hypertension, arrhythmia, uncontrolled hypertension (greater than 140/90 mmHg at screening), tachycardia (resting heart rate > 100 beats per minute); organic epileptic syndrome and active neurological comorbidities; endocrine pathologies (dysthyroidism and adrenals, type I diabetes or insulin-requiring type II diabetes, history of severe hypoglycemia requiring hospitalization); significant impairment of liver function; glaucoma; symptomatic prostatic hypertrophy or bladder neck obstruction; renal failure; respiratory failure; presence of fever or inflammatory syndrome.
* Patient with contraindications to magnetic resonance imaging: patients with a metallic foreign body, pacemaker, neurostimulator or any electronic medical equipment implanted in a non-removable manner, implantable cardiac defibrillators, prostheses, transdermal patches (placed under the skin), catheters (tubes introduced into a vessel or organ), implantable pumps, artificial heart valves, implants to treat deafness.
* Patient at moderate or severe risk of suicide based on clinical judgment (according to the MINI Suicidality Module).
* Patient at high risk of adverse emotional or behavioral reaction based on the investigator's clinical assessment (e.g., severe personality disorder, antisocial behavior, severe current stressors, lack of significant social support, or any psychotic symptoms identified during interviews).

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Activity of the neural circuits responsible for the evaluation of effort before taking psilocybin | Two days before administration of psilocybin
  Brain activity measured by fMRI at resting state and during Effort Expenditure for Rewards Task in the basolateral amygdala, dorsal anterior cingulate cortex, ventral pallidum, ventral striatum and ventral tegmental area
Activity of the neural circuits responsible for the evaluation of effort after taking psilocybin | Five days after administration of psilocybin
  Brain activity measured by fMRI at resting state and during Effort Expenditure for Rewards Task in the basolateral amygdala, dorsal anterior cingulate cortex, ventral pallidum, ventral striatum and ventral tegmental area

SECONDARY OUTCOMES:
Effect of a single-dose administration of psilocybin on self-reported treatment-resistant depression | Day 0
  Quick Inventory of Depressive Symptomatology (QIDS-SR16); 16 items rated from 0 to 3. Total scores range from 0 to 27, with scores of 11 to 15 indicating moderate depression, 16 to 20 reflecting severe depression, and total scores greater than 21 indicating very severe depression.
Effect of a single-dose administration of psilocybin on self-reported treatment-resistant depression | Day 4
  Quick Inventory of Depressive Symptomatology (QIDS-SR16); 16 items rated from 0 to 3. Total scores range from 0 to 27, with scores of 11 to 15 indicating moderate depression, 16 to 20 reflecting severe depression, and total scores greater than 21 indicating very severe depression.
Effect of a single-dose administration of psilocybin on self-reported treatment-resistant depression | Month 1
  Quick Inventory of Depressive Symptomatology (QIDS-SR16); 16 items rated from 0 to 3. Total scores range from 0 to 27, with scores of 11 to 15 indicating moderate depression, 16 to 20 reflecting severe depression, and total scores greater than 21 indicating very severe depression.
Effect of a single-dose administration of psilocybin on self-reported treatment-resistant depression | Month 3
  Quick Inventory of Depressive Symptomatology (QIDS-SR16); 16 items rated from 0 to 3. Total scores range from 0 to 27, with scores of 11 to 15 indicating moderate depression, 16 to 20 reflecting severe depression, and total scores greater than 21 indicating very severe depression.
Effect of a single-dose administration of psilocybin on clinician-rated treatment-resistant depression | Day 0
  Inventory of Depressive Symptomatology, clinician-rated (IDS-C-30); 30 items with each symptom rated from 0 to 3.
Effect of a single-dose administration of psilocybin on clinician-rated treatment-resistant depression | Day 4
  Inventory of Depressive Symptomatology, clinician-rated (IDS-C-30); 30 items with each symptom rated from 0 to 3.
Effect of a single-dose administration of psilocybin on clinician-rated treatment-resistant depression | Month 1
  Inventory of Depressive Symptomatology, clinician-rated (IDS-C-30); 30 items with each symptom rated from 0 to 3.
Effect of a single-dose administration of psilocybin on clinician-rated treatment-resistant depression | Month 3
  Inventory of Depressive Symptomatology, clinician-rated (IDS-C-30); 30 items with each symptom rated from 0 to 3.
Effect of a single-dose administration of psilocybin on anhedonia | Day 0
  Behavioral Activation for Depression Scale (BADS); 9 questions, each rated on a seven-point scale ranging from 0 (not at all) to 6 (completely) for a total score 0-36.
Effect of a single-dose administration of psilocybin on anhedonia | Day 4
  Behavioral Activation for Depression Scale (BADS); 9 questions, each rated on a seven-point scale ranging from 0 (not at all) to 6 (completely) for a total score 0-36.
Effect of a single-dose administration of psilocybin on anhedonia | Month 1
  Behavioral Activation for Depression Scale (BADS); 9 questions, each rated on a seven-point scale ranging from 0 (not at all) to 6 (completely) for a total score 0-36.
Effect of a single-dose administration of psilocybin on anhedonia | Month 3
  Behavioral Activation for Depression Scale (BADS); 9 questions, each rated on a seven-point scale ranging from 0 (not at all) to 6 (completely) for a total score 0-36.
Effect of a single-dose administration of psilocybin on behavioral activation scores | Day 0
  Snaith-Hamilton Pleasure Scale (SHAPS); score ranging from 0-14.
Effect of a single-dose administration of psilocybin on behavioral activation scores | Day 4
  Snaith-Hamilton Pleasure Scale (SHAPS); score ranging from 0-14.
Effect of a single-dose administration of psilocybin on behavioral activation scores | Month 1
  Snaith-Hamilton Pleasure Scale (SHAPS); score ranging from 0-14.
Effect of a single-dose administration of psilocybin on behavioral activation scores | Month 3
  Snaith-Hamilton Pleasure Scale (SHAPS); score ranging from 0-14.
Acceptability of a clinical protocol for psilocybin-assisted therapy in France | Day 4
  SATMED-Q; six dimensions for an overall score from 17 items rated from 0 to 4.
Feasibility of a clinical protocol for psilocybin-assisted in France | Day 4
  Adverse events or tolerance problems collected using the PRISE (Patient Rated Inventory of Side Effect) questionnaire
Effect of psilocybin treatment on states of consciousness. | Day 0
  5-Dimensional Altered States of Consciousness Questionnaire; 94 items rated on a visual analog scale, marked as "no, no more than usual" to "yes, much more than usual", with higher values indicating stronger effects.

CONTACTS AND LOCATIONS:
Overall Officials: Ismaël Conejero, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nîmes, Hôpital Universitaire Carémeau, Nîmes, France